CLINICAL TRIAL: NCT04414917
Title: Reducing Opioid Use/Misuse Through Better Pain Control and Active Pill Dispensing
Brief Title: Reducing Opioid Use and Misuse After Wisdom Molar Extractions
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: iPill Dispenser (Unknown)
Responsible Party: Principal Investigator, Gayathri Dental Subramanian, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2019002739; 1 R21 DA051212-01 (Other: NIH)
Record Dates: First submitted 2020-05-21; First posted 2020-06-04 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pain, Postoperative
Keywords: Impacted third molar extraction; Acute pain management; Active pill dispenser; Opioid misuse reduction
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Prospective randomized blind clinical trial of patients undergoing lower third molar extraction/s to evaluate the ability of the Twin block (local anesthetic nerve block) on side of extraction to reduce post-operative pain and pain medication utilization monitoring with an active pill dispenser
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham injection versus injection of local anesthetic as the Twin block
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Twin Block local anesthetic (Experimental): Patients undergoing extractions of lower wisdom molar/s under intravenous sedation will receive the Twin block local anesthetic (using the standard dental anesthetic 1.8 cc 2% lidocaine with 1:100,000 epinephrine), once, on the side/s of their extraction/s
  Interventions: Drug: Twin block; Device: iPill dispenser
- Control (Sham Comparator): Patients undergoing extractions of lower wisdom molar/s under intravenous sedation will receive the Twin block injection but with no medication administered/dispensed from the syringe, on the side/s of their extraction/s
  Interventions: Device: iPill dispenser

INTERVENTIONS:
Drug: Twin block — Dental local anesthetic administered to target the jaw 'closer' muscles, temporalis and masseter
  Arms: Twin Block local anesthetic
Device: iPill dispenser — An active pill dispenser, regulated by patient's pain score entered on an iPill App installed on their smart phone (iPhone, Android) to dispense opioid (for pain corresponding to severe pain) or prescription strength ibuprofen and acetaminophen (for moderate pain), with over the counter solutions for mild pain recommended. This pill dispenser will be given to all patients, in both Twin block and Control groups, to regulate and monitor their pain experience-driven pain medication regimen. The pill dispenser will be packaged with pain medication (1 dispenser with vicodin, 1 with prescription ibuprofen, 1 with acetaminophen) that has been coencapsulated with ingestible event markers (IEMs, Proteus Discover).
  Other Names: Active pill dispenser

SUMMARY:
Reducing opioid prescription related use and misuse is a major focus for countering the national epidemic of opioid overdose and death. Annually, over 3.5 million predominantly young and healthy individuals undergo outpatient third molar ('wisdom tooth') tooth extractions under sedation and routinely receive postoperative opioid prescriptions. This procedure is among the most prevalent instances of opioid prescriptions dispensed to adolescents, a vulnerable population. This overuse can be minimized by bringing about immediate and sustained pain relief following extractions and by proper monitoring to regulate post-operative opioid usage.

The investigators developed the Twin block, a local anesthetic nerve block that rapidly eases pain from the 'closer' muscles of the jaw and showed its long-term effectiveness in patients with chronic jaw muscle pain. Administering the Twin block immediately following third molar extractions will be an innovative and effective modality to alleviate acute post-procedure pain experienced by the patient and hence reduce the need for post-operative opioid pain medication.

In order to tightly regulate when, how many and to whom the prescribed opioid pill is accessible, this study will utilize the iPill Dispenser®, an active pill dispenser. The iPill device, designated as a Class I 510(k) exempt device by the FDA, includes an App that utilizes biometric user authentication to operate a portable tamper-resistant, pre-calibrated device to regulate, deliver, and monitor opioid usage for pain, preventing overconsumption and diversion. The investigators further plan to 'track' pill swallowing by encapsulating the medication with an ingestible event marker (IEMs, FDA approved Class II device). The hypothesis of this study is that reduction in opioid prescription and its unwarranted use following third molar extractions can be achieved by a combination of Twin block, an active pill dispenser and ingestion tracking. The Specific Aims are:

Specific Aim 1. Compare highest pain after third molar tooth extractions, in patients with and without the twin block.

Specific Aim 2. Compare postoperative opioid consumption during the first 4 days following third molar tooth extractions between patients who got the twin block, with those who do not. Using the iPill dispenser and app and the IEM, the investigators will track opioid consumption for severe pain.

DETAILED DESCRIPTION:
Reducing opioid prescription related use and misuse is a major focus for countering the national epidemic of opioid overdose and death. Annually, over 3.5 million predominantly young and healthy individuals undergo outpatient third molar ('wisdom tooth') tooth extractions and routinely receive postoperative opioid prescription (Moore, Nahouraii et al. 2006). This procedure is among the most prevalent instances of opioid prescriptions dispensed to adolescents and is the subject of a national debate, given the risk for persistent opioid use and abuse in a vulnerable population (Volkow, McLellan et al. 2011, Dowell, Haegerich et al. 2016, Groenewald, Rabbitts et al. 2016, Moore, Dionne et al. 2016, Harbaugh, Nalliah et al. 2018). The investigators believe that this overuse can be minimized by bringing about immediate and sustained pain relief following extractions and by proper monitoring to regulate post-operative opioid usage.

Prolonged mouth opening as well as eccentric and isometric contractions, as are typical during third molar tooth extraction procedures, can result in acute muscle pain in the masticatory or 'chewing' muscles. However, it is common practice to numb only the actual tooth extraction site for postoperative pain management, without evaluating for and addressing acute post-procedure muscle pain. The investigators' preliminary studies have corroborated the efficacy of the Twin block, a local anesthetic, in the diagnosis and management of acute and chronic myogenous orofacial pain stemming from the 'chewing muscles' (Quek, Young et al. 2014, Kanti, Ananthan et al. 2017). The investigators expect that administering the Twin block immediately following third molar extractions, will be an innovative and effective modality to alleviate acute post-procedure pain experienced by the patient and hence reduce the need for post-operative opioid pain medication. Our hypothesis, therefore, is that reduction in opioid prescription and unwarranted use can be achieved by a combination of Twin block and an actively monitored pill dispenser. We have selected the iPill Dispenser® to monitor and regulate post-operative usage.

The iPill device includes an App that utilizes biometric user authentication to operate a portable tamper-resistant, pre-calibrated device to regulate, deliver, and monitor opioid usage for pain, preventing overconsumption and diversion. Coencapsulating the pain pill with the IEM will create a virtual 'time-stamp' by triggering a wireless signal from the IEM, when contacted by stomach acid content, which is detected by a sensor secured on the skin with an adhesive strip.

Therefore, the Specific Aims are:

Specific Aim 1. Compare peak postoperative pain after third molar tooth extractions, with and without the twin block, in a randomized blind prospective clinical study Patients undergoing third molar tooth extractions under 'moderate' (intravenous) sedation, will be randomized to receive either the twin block or a sham injection on the side of their extraction/s. The Twin block and sham injection groups will be compared for peak postoperative pain measured using the numerical pain rating scale (NRS). The investigators predict at least a 50% reduction in percentage of patients reporting significant pain (NRS≥5), in the group randomized to receive the twin block.

Specific Aim 2. Compare postoperative opioid consumption during the first 96 hours following third molar tooth extractions between patients randomized to the control or twin block groups Using the iPill dispenser and app, the investigators will track IEM-co-encapsulated opioid consumption for severe pain among patients randomized to either the sham or Twin block arms. The investigators predict at least a 30% reduction in opioid consumption for severe pain in the group randomized to receive the Twin block. The investigators expect that utilizing the iPill dispenser® and app will enforce rigorous, real-time and accurate monitoring of opioid usage for pain management, overcoming the traditional reliance on patient-reported usage.

POSSIBLE OUTCOMES: This research will potentially transform conventional postoperative pain management following third molar ('wisdom' tooth) extractions. The investigators expect the routine incorporation of the twin block to alleviate post-operative pain, thereby reducing the current reliance on opioid prescriptions in a vulnerable population, especially after a commonplace procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (> 18)
2. American Society of Anesthesiologists Classification I
3. No h/o temporomandibular disorder (TMD) symptoms
4. No h/o trauma to jaws/teeth
5. No h/o surgery in maxillofacial region
6. Presenting for extraction of at least 1 mandibular partially bony/ full bony impacted 'wisdom' or third molar/s under intravenous sedation
7. iPhone or Android smart phone (compatible with iPill® App)
8. Informed consent
9. No cognitive/intellectual disability
10. Not from vulnerable population

Exclusion Criteria:

1. Acute infection or pain in relation to the impacted molars on day of procedure
2. h/o opioid prescription for acute/chronic pain
3. h/o of allergy or contraindication to amide-type local anesthetics, epinephrine or opioids
4. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs)/muscle relaxants/other prescriptions to manage pain/inflammation
5. Refusal/inability to use iPill® App or dispenser
6. h/o eczema

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale score (NRS) | Change in NRS pain scores between baseline and 96 hours post-pain regimen assignment
  Scale from 0 to 10 used to describe no pain (0), mild pain (1-3), moderate (4-6) and severe (7-10) pain. Collection of peak post-procedure, mean, median, quartile pain scores
Pain medication consumed (mg) | Through 96 hours post-procedure
  Dosage of combination opioid, ibuprofen and acetaminophen consumed

SECONDARY OUTCOMES:
Incidence of adverse events | During the first 4 days following procedure
  As described by patients
iPill Dispenser performance- Validation of pills dispensed | During the first 4 days following procedure
  Validation of pills dispensed- correlation between expected and actual number of remaining pills in each dispensers
iPill Dispenser performance- Incidence of dispenser tampering | During the first 4 days following procedure
  Detection of tampering upon inspection of returned dispensers
iPill Dispenser performance- Incidence of failure of operability | During the first 4 days following procedure
  Frequency of failed pill dispensing
iPill Dispenser performance- Percentage of returned dispensers | During the first 4 days following procedure
  Percentage of dispensers returned during post-operative visit
IEM relayed record of pill ingestion | During the first 4 days following procedure
  Log of pills ingested as relayed to IEM App

CONTACTS AND LOCATIONS:
Overall Officials: Gayathri Subramanian, PhD DMD, Principal Investigator — Rutgers School of Dental Medicine; Anayo Adachie, DMD, MD, Principal Investigator — Rutgers School of Dental Medicine
Locations (1):
- Rutgers Health University Dental Associates, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
At this time, we have made the commitment to share aggregate data.(We will consider releasing anonymized individual data upon a case by case documented request that the data is being sought for an appropriate reason).
  With our study design, our basic data will be collected 1. at site of care (dental clinic) and 2. Remotely. Remote data on the app will only be linked with an enrollment number because that data will be collated by our collaborator (Consultant: iPill) and hence will be devoid of identifiers. CRFs will contain data pooled from all the time points in the study and identified only by an enrollment number that will not provide any identifiers. Hence, we will be able to commit to releasing all data collected in this study without compromising patient confidentiality.